CLINICAL TRIAL: NCT03786523
Title: Effects of Time-Restricted Feeding on Nonalcoholic Fatty Liver Disease in Obese Adults: a Randomized Clinical Trial
Brief Title: Time Restricted Feeding on Nonalcoholic Fatty Liver Disease
Acronym: TREATY-FLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2018-160
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Nonalcoholic Fatty Liver Disease; Obesity; Time restricted feeding; Calorie restriction
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Intermittent Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRF (Experimental): Time Restricted Feeding
  Interventions: Behavioral: Time restricted feeding
- CER (Active Comparator): Continuous Energy Restriction
  Interventions: Behavioral: Continuous Energy Restriction

INTERVENTIONS:
Behavioral: Time restricted feeding — Participants will receive a diet of 1500-1800kcal/d for men and 1200-1500kcal/d for women during a window of 8 h/d (8 am to 4 pm).
  Arms: TRF
Behavioral: Continuous Energy Restriction — Participants will follow receive a diet of 1500-1800kcal/d for men and 1200-1500kcal/d for women, without restriction on feeding time.
  Arms: CER

SUMMARY:
Time restricted feeding (TRF) is a novel type of intermittent calorie restriction diet that involves eating a daily period of 8 hours or less. This is a randomized controlled trial to evaluate the effect of time restricted feeding (TRF) on hepatic fat contents and cardiometabolic risk factors in obese adults over 6 months compared to continuous energy restriction (CER).

ELIGIBILITY:
Inclusion Criteria:

1. Man or women aged≥18 years;
2. Subjects with NAFLD determined by MRI (intrahepatic triglyceride content ≥5%);
3. Body mass index (BMI)of 28.0 to 45.0 kg/m2;

Exclusion Criteria:

1. History of alcoholic liver disease, chronic viral hepatitis, drug-induced hepatitis, autoimmune hepatitis, cirrhosis, and liver cancer;
2. History of HIV, or active pulmonary tuberculosis;
3. Diagnosis of type 1 and type 2 diabetes;
4. History of malignant tumors;
5. Serious liver dysfunction or chronic kidney disease (AST or ALT > 3 times the upper limit of normal, or eGFR<30 ml/min/1.73 m2);
6. Significant alcohol consumption in the past six months (Consumed more than 20 g/day for women or 30 g/day for men);
7. History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
8. History of severe gastrointestinal diseases or gastrointestinal surgery in the past 12 months;
9. History of Cushing's syndrome, hypothyroidism, acromegaly, hypothalamic obesity;
10. Being a smoker or having been a smoker in the 3 months prior to their screening visit;
11. Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
12. Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight) ;
13. Women who are pregnant or plan to become pregnant;
14. Patients who cannot be followed for 24 months (due to a health situation or migration);
15. Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Change in intrahepatic fat content | Baseline and months 6
  Intrahepatic fat content will be assessed by MR mDixon-Quant

SECONDARY OUTCOMES:
Change in liver fiber | Baseline and months 6
  Liver fiber will be assessed by liver Fibrotouch
Change in visceral fat | Baseline and months 6
  Visceral fat will be assessed by abdominal CT scan
Change in body fat | Baseline and months 6
  Body fat will be assessed by whole-body dual x-ray system
Change in waist circumference | Baseline and months 6
Change in body weight | Baseline and months 6
Change in HbA1c level | Baseline and months 6
Change in Systolic blood pressure | Baseline and months 6
Change in LDL-c level | Baseline and months 6
Change in serum ALT level | Baseline and months 6
Change in insulin sensitivity | Baseline and months 6
  Insulin sensitivity will be assessed by HOMA-IR
Change in β cell function | Baseline and months 6
  β cell function will be assessed by HOMA-β
Change in pulse wave velocity (PWV) | Baseline and months 6
Depression measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline and months 6
  Scores of PHQ-9
Quality of sleep measured by the Pittsburgh sleep quality index (PSQI) | Baseline and months 6
  Scores of PSQI
Quality of life measured by the 12-item Short-Form Health Survey Questionnaire (SF-12) | Baseline and months 6
  Scores of SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, MD,PhD, Study Chair — Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wei X, Lin B, Huang Y, Yang S, Huang C, Shi L, Liu D, Zhang P, Lin J, Xu B, Guo D, Li C, He H, Liu S, Xue Y, Xu Y, Zhang H. Effects of Time-Restricted Eating on Nonalcoholic Fatty Liver Disease: The TREATY-FLD Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e233513. doi: 10.1001/jamanetworkopen.2023.3513. PMID 36930148